CLINICAL TRIAL: NCT05865327
Title: UltrasouNd-guided Percutaneous Intercostal Nerve Cryoneurolysis for Analgesia Following Traumatic Rib Fracture, a Pilot Randomized Control Trial (UNPIN Trial)
Brief Title: UltrasouNd-guided Percutaneous Intercostal Nerve Cryoneurolysis for Analgesia Following Traumatic Rib Fracture
Acronym: UNPIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5715
Record Dates: First submitted 2023-04-25; First posted 2023-05-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Rib Fractures; Rib Fracture Multiple; Rib; Fracture, With Flail Chest; Pain; Pain, Acute; Pain, Chronic; Trauma; Trauma Injury
Keywords: Cryoneurolysis; Rib Fracture Pain; Intercostal Nerve Block
MeSH Terms: conditions — Rib Fractures; Fractures, Bone; Pain; Acute Pain; Chronic Pain; Wounds and Injuries; Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, parallel, randomized, blinded (participant, data collectors/analysts) pilot feasibility trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the anesthesiologist responsible for performing cryoneurolysis will be aware of group allocation. All others, including participants, other clinical team, data collectors and analysts will be blinded. Participants in the control group will receive sham cryoneurolysis to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoneurolysis Group (Experimental): In addition to all standard of care analgesia treatments, CN will be performed on the ICN of each broken rib using the Iovera CN device and Generation 2 Iovera tip under ultrasound guidance.
  Interventions: Procedure: Cryoneurolysis
- Standard Care Group (Sham Comparator): Participants in the control group will receive all standard of care analgesia treatments as well as sham CN (i.e., application of device without skin puncture or activation of unit) to maintain participant blinding.
  Interventions: Procedure: Sham Cryoneurolysis

INTERVENTIONS:
Procedure: Cryoneurolysis — Cryoneurolysis will be performed on the intercostal nerve associated with each fractured rib using a handheld cryoneurolysis machine (Iovera). Cryoneurolysis will consist of two 103 second cycles (includes cooling, ice ball formation and warming time) per rib fracture level. Ultrasound guidance will be used to identify appropriate rib fracture levels and to target the device tip in real time. All participants will also receive standard multimodal analgesia and ESP catheter infusion.
  Arms: Cryoneurolysis Group
Procedure: Sham Cryoneurolysis — Participants in the control group will receive sham CN (i.e., application of device without skin puncture or activation of unit) to maintain participant blinding. All participants will also receive standard multimodal analgesia and ESP catheter infusion.
  Arms: Standard Care Group

SUMMARY:
Traumatic rib fractures (i.e., broken ribs caused by a physical injury) are common and very painful. They also often lead to serious complications, more time spent in hospital, and can even lead to death. Even after rib fractures have healed, they can lead to long-term pain and a lower quality of life.

A technology called cryoneurolysis, which acts to freeze nerves causing pain using a small tool which can turn very cold, is a promising new way to manage rib fracture pain. This study is a test with a small number of people to see if it is feasible to use this technology for patients with rib fractures. If this is successful, we will recruit more people for a larger study to see if cryoneurolysis, along with standard pain control techniques, is better at stopping pain, compared to just the normal techniques alone. Participants in our study will be asked to rate their pain, and record pain medications that they take for 3 months after their pain procedure.

DETAILED DESCRIPTION:
More than 100,000 people a year suffer from traumatic rib fractures. Pain from rib fractures impairs the ability to inspire deeply and cough effectively, predisposing patients to severe, potentially life threatening complications and increased healthcare costs. For many patients, this pain can also persist long after the acute injury has healed, delaying recovery and reducing quality of life.

Current pain interventions, including multimodal analgesia and local anesthetic-based nerve blocks, are useful, but are limited by a short duration of effectiveness, and/or risk of complications. Cryoneurolysis (CN) is a new method to control pain which acts to freeze intercostal nerves (ICNs) associated with fractured ribs using a handheld device. This freezing action causes neurons to undergo Wallerian degeneration distally from the site of ablation and thus exhibit an extended but reversible block.

This study is a single-site, randomized, pilot study to assess the feasibility of recruitment, randomization, and protocol adherence of providing cryoneurolysis for patients with traumatic rib fractures. Secondary data from the pilot trial designed to assess the effectiveness of the intervention (pain scores, opioid usage, etc.) will be included in the analysis of the full trial if feasible. The objective of the full trial is to demonstrate that cryoneurolysis of ICN, in addition to standard analgesic practice, provides superior, prolonged analgesia.

Participants (individuals aged 18-85, with 3-8 unilateral traumatic rib fractures) will be randomized 1:1 in blocks of 4, stratified by number of rib fractures (> 4 or ≤4) and the presence/absence of flail segment, to receive the current standard of practice for rib fractures (multimodal analgesia and erector spinae plane (ESP) catheter infusion) with or without the addition of CN. Participants in the standard care group will receive a sham CN procedure to maintain blinding.

All participants (both groups) will receive standard of care analgesia. Specifically, an ultrasound-guided ESP catheter will be placed as per standard protocols. 20cc of 0.5% ropivacaine and 1% lidocaine will be injected through the catheter, followed by a basal infusion of 2 cc/hr of 0.2% ropivacaine (to maintain catheter patency) with an on demand patient controlled regional anesthesia (PCRA) dose of 10cc 0.2% ropivacaine available hourly until patient has met criteria for APS discharge or pain is controlled such that PCRA use is < 2 boluses over 12 hrs and NRS < 3 with deep breathing and coughing.

Standard multimodal analgesia including Tylenol 1000mg QID, Celebrex 200mg BID (or ketorolac 7.5 QID), Pregabalin 50mg BID, and/or PRN oral hydromorphone (1-4mg) will also be provided. Additional analgesics include intravenous ketamine at a dose of 0.1-0.2 mg/kg/hr of lean body weight in the event of consistent NRS pain scores > 6, and up to 0.05 mg/kg of intravenous midazolam for anxiolysis and 1mcg/kg of intravenous fentanyl for comfort during positioning, as required.

Participants will remain in the study for 3 months from the date of the block procedure. They will be followed daily while in hospital and using a pain diary following discharge (weekly pain scores and daily opioid usage). Additionally, follow-ups will be completed at 1h, 24h, 48h, 1 week, 1 month, and 3 months post block procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Unilateral traumatic rib fractures (3 to 8)
* Candidate for ESP block catheter
* Within 48hrs of admission to hospital

Exclusion Criteria:

* Lack of patient consent; unlikely to comply with follow up
* Unable to use Patient Controlled Regional Analgesia (Ventilated/sedated patients or Moderate to severe traumatic brain injury)
* Chronic pain (opioid use > 30mg oral morphine equivalent per day)
* Substance use disorder
* CrCl < 50
* BMI > 45
* Significant distracting injuries (unreduced long bone fractures, unstable pelvic or spine fractures and patients requiring trauma laparotomy- also preclude positioning for block placement (lateral decubitus or sitting up))
* Contraindications for ESP catheter placement (pre-existing medical/neurological/hematologic diseases, localized infection/trauma at site of intervention, allergy to amide local anesthetics)
* Contraindications to CN (cryoglobulinemia, paroxysmal cold hemoglobinuria, multiple myeloma and cold urticarial).
* Unable to return to Trauma Recovery Clinic (in-person or virtual) at 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants randomized over an 8 month period | Entire pilot study (approximately 8 months)
  Goal of 3 participants per month for 8 months
Number of participants able to adhere to the protocol | Entire pilot study (approximately 8 months + 3 month follow-up)
  Goal of > 90%
Number of participants able to adhere to the follow-up | 3 month follow-up
  Goal of > 90%
Rate of Adverse events | 3 month follow-up
  Ensure no adverse events (short or long term) associated with CN

SECONDARY OUTCOMES:
Pain Severity during deep inspiration 24 hours post ESP catheter placement | 24 hours post placement of ESP catheter
  Pain measured using Numeric Pain Rating Scale
Time to discontinuation of ESP catheter | Until ESP catheter removal (usually < 7 days)
  Based on when patient has met criteria for APS discharge or pain is controlled such that PCRA use is < 2 boluses over 12 hrs and NRS < 3 with deep breathing and coughing
ESP catheter use | Until ESP catheter removal (usually < 7 days)
  Cumulative volume of local anesthetic solution used via ESP catheter patient controlled reginal analgesia
Opioid consumption in hospital and after discharge | Daily for 90 days after block placement
  Determined from medical records (in-hospital) and via a daily pain diary (post-discharge). Calculated in Oral Morphine Equivalents.
Pain Intensity at 1 and 3 months | 1 and 3 month follow-ups
  As measured using Numeric Pain Rating Scale (0-10) , at rest and during deep inspiration
Oxygen requirements | Pre-intervention, post intervention, then daily until discharge
  Room air oxygen saturation (SpO2) and requirement for supplementary O2 to maintain SpO2 > 92%
Pulmonary Function Testing | Pre-intervention, post intervention, then daily until discharge
  FVC
Pulmonary Function Testing | Pre-intervention, post intervention, then daily until discharge
  FEV1
Pulmonary Function Testing | Pre-intervention, post intervention, then daily until discharge
  Peak Inspiratory flow
Pulmonary Function Testing | Pre-intervention, post intervention, then daily until discharge
  Peak Expiratory Flow
Length of Stay in hospital | Date of admission to date discharge
  Hospital discharge date
Length of Stay on acute pain service (APS) | Date of admission to date of discharge from acute pain service
  Criteria include on oral meds without continuous regional analgesia or intravenous opioids
Time to achieve discharge criteria for isolated chest injury | Date of admission until discharge criteria met
  Criteria include on oral meds without continuous regional analgesia, chest tube out and chest well evacuated (e.g. no evidence of retained hemothorax), and no supplemental O2
Patient satisfaction | 48 post block procedure, and 1 week, 1 month and 3 month follow-ups
  Patient satisfaction assessed using Patients' Global Impression of Change (PGIC) scale
Incidence of chronic rib fracture pain | 3 month follow-up
  As assessed using Brief Pain Inventory (BPI) questionnaire
Adverse events | until 3 month follow-up
  Adverse events to be recorded include: local anesthetic complications, catheter related complications (clotting, migration), procedural complications (pneumothorax, bleeding, infection), and neurological disturbances (dysesthesia, hyperalgesia, allodynia) in area of rib fracture

OTHER OUTCOMES:
Pain Intensity | 1h and 48h, post block placement, daily in hospital, weekly post discharge and at 1 week follow-up
  As measured using NRS-11, at rest and during deep inspiration

CONTACTS AND LOCATIONS:
Overall Officials: Ben Safa, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available upon reasonable request to study PI following publication of full trial results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This is a pilot trial and full inferential analysis will not be conducted until completion of the full trial. As such, data will be available following publication of the primary results of the subsequent full trial.
Access Criteria: Data and supporting information will be made available following reasonable request directly to study PI.